CLINICAL TRIAL: NCT06578819
Title: Evaluating the Impact of Doll Therapy on Agitation, Nutritional Status, and Activities of Daily Living in Agitated Older Adults With Dementia: A Randomized Controlled Trial
Brief Title: Doll Therapy for Agitated Elderly Dementia People
Acronym: DT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, AYNUR CİN, Principal investigator, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25/10/2023 date and 2023/5
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Agitation
Keywords: dementia; doll therapy; nursing; daily activity; nutrition
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: pre-test and post-test case control
Who Masked: Outcomes Assessor
Masking Description: Due to the inherent nature of doll therapy, blinding of participants and the researcher administering the intervention was not feasible. Participants were aware if they were receiving doll therapy, and the researcher delivering the therapy was also aware of the assigned group. However, to minimize detection bias, all outcome assessors who administered the CMAI, EdFED, and Katz ADL were rigorously blinded to group allocation. These assessors were specifically instructed not to inquire about or discuss the participants' treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- experimental group (moderate dementia) (Experimental): Prior to the start of the study, the MMSE was administered to identify patients in the experimental group with severe and moderate dementia. Patients who scored between 0 and 17 on the MMSE were classified as having severe dementia, while those who scored between 18 and 23 were classified as having moderate dementia and included in the study. Before the intervention began, the vital signs of elderly patients with dementia were recorded and documented using the Structured Patient Information Form.
  Toy doll therapy was administered by the same researcher to elderly dementia patients who scored 35 or higher on the long form of the CMAI. In accordance with the principles of toy doll therapy as outlined in the literature, the intervention was conducted four days per week over a total period of 12 weeks for agitated elderly patients with dementia.
  Three standardized assessment tools were administered to both the moderate and severe dementia groups at three time point
  Interventions: Behavioral: doll therapy
- control group (moderate dementia) (No Intervention): Before the study commenced, the MMSE was administered to identify patients in the control group with moderate and severe dementia. Patients scoring between 0 and 17 were classified as having severe dementia, while those scoring between 18 and 23 were classified as having moderate dementia and included in the study. Prior to the start of the intervention, the vital signs of elderly patients with dementia were recorded and documented using the Structured Patient Information Form.
  Elderly dementia patients who scored above 35 on the long form of the CMAI were included in the control group. No intervention was administered to either subgroup (moderate and severe dementia patients) in the control group. These patients continued to receive their routine medical care and treatment.
  Patients in the control group were assessed using the CMAI, the EdFED, and the Katz ADL at three time points: at the beginning of the study, at the midpoint (week 6), and at the end (week 12).
- experimental group (severe dementia) (Experimental): Prior to the start of the study, the MMSE was administered to identify patients in the experimental group with severe and moderate dementia. Patients who scored between 0 and 17 on the MMSE were classified as having severe dementia, while those who scored between 18 and 23 were classified as having moderate dementia and included in the study. Before the intervention began, the vital signs of elderly patients with dementia were recorded and documented using the Structured Patient Information Form.
  Toy doll therapy was administered by the same researcher to elderly dementia patients who scored 35 or higher on the long form of the CMAI. In accordance with the principles of toy doll therapy as outlined in the literature, the intervention was conducted four days per week over a total period of 12 weeks for agitated elderly patients with dementia.
  Three standardized assessment tools were administered to both the moderate and severe dementia groups at three time point
  Interventions: Behavioral: doll therapy
- control group (severe dementia) (No Intervention): Before the study commenced, the MMSE was administered to identify patients in the control group with moderate and severe dementia. Patients scoring between 0 and 17 were classified as having severe dementia, while those scoring between 18 and 23 were classified as having moderate dementia and included in the study. Prior to the start of the intervention, the vital signs of elderly patients with dementia were recorded and documented using the Structured Patient Information Form.
  Elderly dementia patients who scored above 35 on the long form of the CMAI were included in the control group. No intervention was administered to either subgroup (moderate and severe dementia patients) in the control group. These patients continued to receive their routine medical care and treatment.
  Patients in the control group were assessed using the CMAI, the EdFED, and the Katz ADL at three time points: at the beginning of the study, at the midpoint (week 6), and at the end (week 12).

INTERVENTIONS:
Behavioral: doll therapy — Doll therapy applied to the experimental group 4 days a week.
  Arms: experimental group (moderate dementia); experimental group (severe dementia)

SUMMARY:
This study is designed to determine the effect of doll therapy on the levels of agitation, nutrition, and daily living activities in elderly patients with dementia and agitation.

DETAILED DESCRIPTION:
Elderly patients with agitation and dementia incur significant costs for healthcare services. Additionally, it is known that agitation can impose a burden on caregivers and has the potential to cause harm to the individual and those around them. This study is planned to determine the effect of doll therapy on the levels of agitation, nutrition, and daily living activities in elderly patients with dementia and agitation.

ELIGIBILITY:
Inclusion Criteria:

Aged 65 years or older, met the DSM-IV diagnostic criteria for dementia, clinical diagnosis of Alzheimer's disease, diagnosis of dementia (moderate or severe) confirmed by a neurologist, must be able to swallow tablets, had sufficient hand motor skills to hold and care for a doll, had adequate visual acuity to recognize the doll, had no significant communication impairments, were personally willing to participate in the study, had the consent of their legal guardians or family members for participation in the study. Exhibiting agitation, defined as a score of 35 or higher on the long form of the CMAI.

Exclusion Criteria:

Participants were excluded from the study if they had a diagnosis of mild dementia, were experiencing an acute exacerbation of a systemic illness, or had a diagnosed psychological disorder, Insulin dependent diabetes and thyroid disease. Additionally, elderly individuals who experienced difficulty accepting and forming a relationship with the doll after two attempts were excluded from the study. Those who initially accepted the doll but later abandoned it were also excluded. Lastly, participants who reported that the doll triggered negative associations or adverse emotional responses were excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
The Edinburgh feeding evaluation in dementia (EdFED) scale (Nutrition) | 12 week
  One standardized assessment tool administered to both the moderate and severe dementia groups at three time points: at the beginning of the study, at the midpoint (week 6), and at the end (week 12). These tool included the EdFED. The scale consists of 11 items and can be administered in less than five minutes. The first 10 items address feeding behaviors during meals; each item is scored based on the frequency of occurrence. If the behavior does not occur during meals, it is scored as "never" (0 points), if it occurs 2-3 times a week it is scored as "sometimes" (1 point), and if it occurs more than 4 times a week, it is scored as "often" (2 points). There is no cutoff score or reverse scoring in the scale. The total score obtained from the first 10 items ranges from 0 to 20, with a score of 20 indicating the most severe condition. The total score can be used to track changes in the patient's nutritional status. The level of support the patient requires is determined by item 11.
Cohen-Mansfield Agitation Inventory (Agitation) | 12 week
  One standardized assessment tool administered to both the moderate and severe dementia groups at three time points: at the beginning of the study, at the midpoint (week 6), and at the end (week 12). These tool included the CMAI. The CMAI uses a Likert scale, where each item is scored from "1 never" to "7 several times per hour." The total score is calculated based on a maximum of 32 items, with a possible total score range from 29 to 181.
Katz Daily Life Activities Scale (Daily activities) | 12 week
  One standardized assessment tool administered to both the moderate and severe dementia groups at three time points: at the beginning of the study, at the midpoint (week 6), and at the end (week 12). These tool included the Katz ADL. The scale assigns scores to daily activities such as bathing, dressing, toileting, mobility, continence, and feeding. Based on the total score, the individual's level of dependence is classified as follows: 0-6 points indicate dependence, 7-12 points indicate partial dependence, and 13-18 points indicate independence. Each item on the Katz ADL scale includes response options indicating whether the individual is independent, partially dependent, or dependent. The scale assesses six fundamental activities: bathing, dressing, toileting, transferring, continence, and feeding.

SECONDARY OUTCOMES:
The Edinburgh feeding evaluation in dementia (EdFED) scale (Nutrition) | 12 week
  One standardized assessment tool administered to both the moderate and severe dementia groups at three time points: at the beginning of the study, at the midpoint (week 6), and at the end (week 12). These tool included the EdFED. The scale consists of 11 items and can be administered in less than five minutes. The first 10 items address feeding behaviors during meals; each item is scored based on the frequency of occurrence. If the behavior does not occur during meals, it is scored as "never" (0 points), if it occurs 2-3 times a week it is scored as "sometimes" (1 point), and if it occurs more than 4 times a week, it is scored as "often" (2 points). There is no cutoff score or reverse scoring in the scale. The total score obtained from the first 10 items ranges from 0 to 20, with a score of 20 indicating the most severe condition. The total score can be used to track changes in the patient's nutritional status. The level of support the patient requires is determined by item 11.
Cohen-Mansfield Agitation Inventory (Agitation) | 12 week
  One standardized assessment tool administered to both the moderate and severe dementia groups at three time points: at the beginning of the study, at the midpoint (week 6), and at the end (week 12). These tool included the CMAI. The CMAI uses a Likert scale, where each item is scored from "1 never" to "7 several times per hour." The total score is calculated based on a maximum of 32 items, with a possible total score range from 29 to 181.
Katz Daily Life Activities Scale (Daily activities) | 12 week
  One standardized assessment tool administered to both the moderate and severe dementia groups at three time points: at the beginning of the study, at the midpoint (week 6), and at the end (week 12). These tool included the Katz ADL. The scale assigns scores to daily activities such as bathing, dressing, toileting, mobility, continence, and feeding. Based on the total score, the individual's level of dependence is classified as follows: 0-6 points indicate dependence, 7-12 points indicate partial dependence, and 13-18 points indicate independence. Each item on the Katz ADL scale includes response options indicating whether the individual is independent, partially dependent, or dependent. The scale assesses six fundamental activities: bathing, dressing, toileting, transferring, continence, and feeding.

CONTACTS AND LOCATIONS:
Overall Officials: AYNUR CIN, DR, Study Director — Gümüşhane Universıty
Locations (1):
- Kelkit State Hospital, Kelkit, Gümüşhane Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
STUDY PROTOCOL
Supporting Information: Study Protocol
Time Frame: 15 DECEMBER 2024 -31 MAY 2024
Access Criteria: ACCESS WILL BE PROVIDED WITHIN THE SCOPE OF THE RESEARCHER'S PERMISSION